CLINICAL TRIAL: NCT01440478
Title: Impact of Variations in Urinary pH on the Pharmacokinetics of LY2140023 and LY404039 in Healthy Subjects
Brief Title: The Effects of Urinary pH Changes on an Investigational Compound in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 12322; H8Y-EW-HBBX (Other: Eli Lilly and Company); 2011-003215-36 (Registry Identifier: EuDraCT)
Record Dates: First submitted 2011-08-31; First posted 2011-09-26 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — LY 2140023; Ammonium Chloride; Sodium Bicarbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LY2140023 + ammonium chloride (Experimental): 1 g of ammonium chloride administered orally every 3 hours for 33 hours (totaling 12 doses) in combination with a single 80 mg dose of LY2140023 administered orally 17 hours after first dose of ammonium chloride (acidified urine). All participants will receive the three treatments in a randomized order. There will be a minimum of a 5 day wash out period between treatment periods.
  Interventions: Drug: LY2140023; Drug: Ammonium chloride
- LY2140023 + sodium bicarbonate (Experimental): 4 g of sodium bicarbonate administered orally every 4 hours for 32 hours (totaling 9 doses) in combination with a single 80 mg dose of LY2140023 administered orally 18 hours after first dose of sodium bicarbonate (alkalized urine). All participants will receive the three treatments in a randomized order. There will be a minimum of a 5 day wash out period between treatment periods.
  Interventions: Drug: LY2140023; Drug: Sodium bicarbonate
- LY2140023 (Experimental): A single 80 mg dose of LY2140023 administered orally (normal urine). All participants will receive the three treatments in a randomized order. There will be a minimum of a 5 day wash out period between treatment periods.
  Interventions: Drug: LY2140023

INTERVENTIONS:
Drug: LY2140023 — Administered orally
Drug: Ammonium chloride — Administered orally
  Arms: LY2140023 + ammonium chloride
Drug: Sodium bicarbonate — Administered orally
  Arms: LY2140023 + sodium bicarbonate

SUMMARY:
This study is designed to explore the effect of increased and decreased urinary pH on the single pharmacokinetic (PK) dose of LY2140023 and its active metabolite LY404039. All participants will receive the three treatments in a randomized order.

ELIGIBILITY:
Inclusion Criteria:

* are overtly healthy males or females, as determined by medical history and physical examination
* female subjects of childbearing potential, who test negative for pregnancy at screening. Male subjects/female subjects of childbearing potential/female subjects who have been sterilized by tubal ligation and their partners will be required to use a condom (male condom or female condom) used in conjunction with spermicidal gel, foam, cream, film, or suppository from the time of screening (female subjects) or dosing (male subjects) until 3 months after the last dose of investigational product. Male subjects with female partners of childbearing potential and female subjects of childbearing potential will be requested to use an additional highly effective form of contraception from the first dosing occasion until 3 months after the last dose of investigational product. The additional method of contraception can be any of the following: diaphragm or cervical vault cap used in conjunction with spermicidal gel, foam, cream, film, or suppository; male sterilization, with the appropriate post vasectomy documentation of the absence of sperm in the ejaculate, or for female subjects the vasectomized male partner should be the sole partner for that subject; true abstinence (this must be due to subject's lifestyle choice; placement of an effective hormonal intrauterine device (IUD) (i.e. Mirena Coil) (steel or copper IUDs are not acceptable); or established use of oral, injected, or implanted hormonal methods of contraception
* female subjects who are of non childbearing potential i.e. post menopausal or permanently sterile following hysterectomy, bilateral salpingectomy or confirmed tubal occlusion (not tubal ligation). Postmenopausal is defined as at least 1 year post cessation of menses (without an alternative medical cause) with follicle stimulating hormone (FSH) ≥40 mIU/mL
* have a body mass index (BMI) of 19 to 32 kg/m^2, inclusive, at the time of screening
* have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* have venous access sufficient to allow for blood sampling
* are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* have given written informed consent approved by Lilly and the chosen ethical review board (ERB)
* are willing to adhere to dietary requirements

Exclusion Criteria:

* are currently enrolled in, have completed or discontinued within the last 90 days from, a clinical trial involving an investigational product; or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* have known allergies to LY2140023, LY404039, ammonium chloride, sodium bicarbonate, related compounds, or any components of the formulation
* are persons who have previously received the investigational product in this study, withdrawn from this study or any other study investigating LY2140023 or LY404039
* have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* have an abnormality in the serum chemistry of calcium, sodium, magnesium, or potassium, that, in the opinion of the investigator, increases the risks associated with participating in the study
* have an abnormal supine and standing blood pressure or pulse rate, as determined by the investigator
* have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* have evidence of significant active neuropsychiatric disease (for example, manic depressive illness, schizophrenia, depression)
* have increased risk of seizures based on a history of:

  * one or more seizures (except for a single simple febrile seizure [lacking focality and lasting less than 15 minutes, not associated with a central nervous system (CNS) infection or severe metabolic disturbance] as a child between ages 6 months to 5 years)
  * head trauma with loss of consciousness or a post concussive syndrome within 1 year or lifetime history of head trauma with persistent neurological deficit (focal or diffuse)
  * CNS infection, uncontrolled migraine or transient ischemic attack (TIA) within 1 year; stroke with persistent neurological deficit (focal or diffuse), uncontrolled migraine is defined as migraine attacks that produce headache lasting up to 72 hours and are often accompanied by associated symptoms (nausea, photophobia, and phonophobia) that impair well-being and disrupt social functioning. TIA is defined as "mini-stroke" caused by temporary disturbance of blood supply to an area of the brain, which results in a sudden, brief decrease in brain function
  * CNS infection with persistent neurological deficit (focal or diffuse)
  * brain surgery
  * electroencephalogram (EEG) with paroxysmal (epileptiform) activity (isolated spikes waves, repetitive bursts of sharp waves, paroxysmal activity, frank seizures, spike-wave complexes, or sharp-slow wave complexes, or as locally defined)
  * brain structural lesion, including developmental abnormalities, as determined by examination or imaging studies (does not include hydrocephalus unless treated by shunt or resulting in neurological deficits)
* show evidence of known substance dependence or abuse within 6 months prior to the study (according to Diagnostic and Statistical Manual of Mental Disorders [DSM IV] diagnosis), or regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* show evidence of hepatitis C and/or positive hepatitis C antibody
* show evidence of hepatitis B and/or positive hepatitis B surface antigen
* are women with a positive pregnancy test or women who are lactating
* intend to use over the counter (excluding most vitamin/mineral supplements but including herbal remedies/health supplements or prescription medication (excluding paracetamol, oral contraceptives and hormone replacement therapy) within 14 days prior to dosing of LY2140023. If this situation arises, inclusion of an otherwise suitable subject may be at the discretion of the investigator in consultation with the Lilly Clinical Pharmacologist (CP) or designee
* have donated blood of more than 500 mL within 3 months prior to screening
* have an average weekly alcohol intake that exceeds 28 units per week (males up to age 65) and 21 units per week (females), or are unwilling to stop alcohol consumption for the duration of the study (1 unit equals 12 oz or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* have a clinical significant abnormality in the neurological examination
* subjects judged prior to randomization to be at suicidal risk by the investigator
* subjects who are unwilling to refrain from tobacco or nicotine containing products while in the Clinical Research Unit (CRU) or are unable to abide by the CRU restrictions
* history of, in the opinion of the investigator, excessive methylxanthine use within previous 6 months, such as >6 cups of coffee (or equivalent) per day
* show evidence of active renal disease (for example, diabetic renal disease, polycystic kidney disease) or creatinine clearance (CrCL) less than 80 mL/min (as calculated by the Cockcroft Gault equation) Men: [(140 - age) * (weight in kg) * 1.23] / (serum creatinine in µmol/L). Women: [(140 - age) * (weight in kg) * 1.04] / (serum creatinine in µmol/L)
* show evidence of pruritus or skin exfoliation
* have an eosinophil count >1.5 x 109/L
* have creatine kinase (CK) >5 x upper limit of normal (ULN)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: area under the concentration versus time curve (AUC) of LY2140023 and LY404039 | Predose and up to 24 hours post dose after LY2140023 dosing for each of the 3 treatment periods
Pharmacokinetics: maximum observed drug concentration (Cmax) of LY2140023 and LY404039 | Predose and up to 24 hours post dose after LY2140023 dosing for each of the 3 treatment periods
Change from baseline in urine pH | Predose and up to 24 hours post dose after LY2140023 dosing for each of the 3 treatment periods

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559), Mon - Fri, from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Leeds, United Kingdom